CLINICAL TRIAL: NCT02099812
Title: Web-based Collection of Data on Obesity and Health Behavior
Status: Completed | Type: Observational
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jeffrey Stein, Professor, Virginia Polytechnic Institute and State University
Other Study IDs: VT-12-483
Record Dates: First submitted 2014-03-10; First posted 2014-03-31 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese: Obese individuals
- Non-obese: Non-obese individuals

SUMMARY:
Low socioeconomic status (low SES), as defined by educational attainment and income, has been associated with obesity in industrialized nations. Low SES has been related to impulsive decision-making characterized by steep devaluation of future outcomes (delay discounting, DD) and a greater motivation to obtain food (food reinforcement, FR). DD and FR have been shown to interactively predict ad libitum energy intake in laboratory studies, such that participants exhibiting high FR as well as high DD consume the most food. Obesity often results from energy intake in excess of physiologic needs, and thus a plausible mechanism is that low SES environments increase FR and DD, leading to overeating and obesity. The primary aims of this study are to determine whether FR and DD interact to predict BMI, and whether differences in FR and DD mediate the relationship between low SES and obesity, in a large sample of US adults of varying BMI. In addition, whether high FR and high DD are related to unhealthy food purchasing and eating behaviors will be assessed. It is anticipated that high FR and DD will be related to unhealthy food purchasing and eating behaviors.

DETAILED DESCRIPTION:
In this study potential participants who log in to the Amazon Mechanical Turk website as a worker and who have a HIT approval rate of at least 90% will be allowed to view and participate in the study. If a potential participant agrees to participate in the study by accepting the HIT, the participant will be asked to complete a brief survey (approximately 150 questions; see sample survey in "other supporting documents") and various decision making tasks (e.g., delay discounting assessment, reinforcer valuation assessment etc.). This survey and accompanying tasks will solicit: (a) general demographic information such as gender, age, income, and education; (b) information about their health and health behavior practices, such as eating habits, alcohol and cigarette use; (c) questions about their food preferences and value of foods; (d) information about their valuation of immediate versus distant events/rewards.

ELIGIBILITY:
Inclusion Criteria:

* Be a registered Amazon Mechanical Turk user.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Amazon Mechanical Turk users
Sampling Method: Non-Probability Sample
Enrollment: 1585 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Delay discounting rate | 1 hour
  Degree to which future rewards are devalued
Food reinforcement | 1 hour
  Participant's valuation of food items.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Epstein LH, Jankowiak N, Lin H, Paluch R, Koffarnus MN, Bickel WK. No food for thought: moderating effects of delay discounting and future time perspective on the relation between income and food insecurity. Am J Clin Nutr. 2014 Sep;100(3):884-90. doi: 10.3945/ajcn.113.079772. Epub 2014 Jul 9. PMID 25008855